CLINICAL TRIAL: NCT04529330
Title: Acute Compartment Syndrome
Brief Title: The Research About Acute Compartment Syndrome
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HZY001ACS
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Acute Compartment Syndrome
Keywords: ACS; Tibial plateau fractures; Tibial shaft fractures
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Fasciotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fractures with blister appeared: tibial plateau fractures with blister observed
  Interventions: Procedure: fasciotomy
- fractures without blister appeared: tibial plateau fractures without blister observed
  Interventions: Procedure: fasciotomy

INTERVENTIONS:
Procedure: fasciotomy — if it was suspected with ACS, the fasciotomy was conducted. but if the blister observed, it means decreased conmpartment sydrome. therefore, the blister observed can avoid unnecessary fasciotomy to patients suspected with ACS

SUMMARY:
Acute compartment syndrome (ACS) is defined as a clinical entity originated from trauma or other conditions, and remains challenging to diagnose and treat effectively. Threre is the controversy in diagnosing, treating ACS. It was found that there was no criterion about the ACS, and result unnecessary osteotomy. The presence of clinical assessment (5P) always means the necrosis of muscles and was the most serious or irreversible stage of ACS. Besides pressure methods, the threshold of pressure identifying ACS was also controversial.

ELIGIBILITY:
Inclusion Criteria:

* Fracture patients with Schatzker V and VI,
* Who were older than eighteen years.

Exclusion Criteria:

* The exclusion criteria were pathologic, extra-articular proximal tibial fracture,
* Patients who was eighteen years or younger.
* Patients treated with other implant,
* underwent conservative management were also excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The severe tibial plateau (Ⅴand Ⅵ according to Schatzker's classification) in our hospital who will be treated with open internal fixation in our hospital
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-09-09 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
injury mechanism | up to 1 weeks
  The relative data was collected about injury mechanism such as high falling accident, traffic accident, fall from standing height,Crushing
the time when the blister appeared | up to 4 weeks
  The relative data was collected about the time when the blister appeared after injury
time to reconstructive surgery | time to when the surgery was conducted after 2 weeks
  The relative data was collected about time to reconstructive surgery
union time | through study completion, an average of 1 year
  The relative data was collected about union time
No non-anatomic gap or step (larger than 5 mm) | through study completion, an average of 1 year
  The relative data was collected about complications
secondary loss of reduction | through study completion, an average of 1 year
  The relative data was collected about complications
Deep venous thrombosis | through study completion, an average of 1 year
  The relative data was collected about complications
superficial wound problems | through study completion, an average of 1 year
  The relative data was collected about complications
blister skin immunochemistry and immunofluorescence analysis | through study completion, an average of 1 year
  CK1, 5, 10, claudin 1, 2 and occludin as determined by immunochemistry analysis, and skin barrier proteins; claudin 1, 2 and occludin was determined by immunofluorescence analysis and qPCR.

SECONDARY OUTCOMES:
CK levels | through hospitalization completion, an average of 1 month
  CK levels
chloride levels | through hospitalization completion, an average of 1 month
  chloride levels
UREA levels | through hospitalization completion, an average of 1 month
  UREA levels

OTHER OUTCOMES:
LKS score | through study completion, an average of 1 year
  Lysholm knee score
VAS scores | through study completion, an average of 1 year
  visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Hou Zhiyong, Doctor, Principal Investigator — Hebei Medical University Third Hospital
Locations (1):
- the Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
acute compartment syndrome
Supporting Information: Study Protocol
Time Frame: 2 years after the experiment was conducted
Access Criteria: all authors focusing on ACS research

REFERENCES:
- [Background] Guo J, Yin Y, Jin L, Zhang R, Hou Z, Zhang Y. Acute compartment syndrome: Cause, diagnosis, and new viewpoint. Medicine (Baltimore). 2019 Jul;98(27):e16260. doi: 10.1097/MD.0000000000016260. PMID 31277147
- [Derived] Wang T, Yang S, Guo J, Long Y, Hou Z. Predictors of muscle necrosis in patients with acute compartment syndrome. Int Orthop. 2023 Apr;47(4):905-913. doi: 10.1007/s00264-023-05699-9. Epub 2023 Jan 30. PMID 36715712